CLINICAL TRIAL: NCT07073001
Title: UMG-CHUSE Study: Three-month Follow-up Analysis of Social Recommendations Issued by the Mobile Geriatric Team.
Brief Title: Three-month Follow-up Analysis of Social Recommendations Issued by the Mobile Geriatric Team
Acronym: UMG-CHUSE
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN692025/CHUSTE
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Geriatric; Care Coordination; Readmission, Hospital
Keywords: Geriatrics; Mobile Geriatric Team; Care coordination; Social recommandations; Elderly care; Hospital readmission
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients included: Patients aged 75 and over who have been assessed by the CHUSE mobile geriatrics team and have received social recommendations.
  Interventions: Other: Telephone interview

INTERVENTIONS:
Other: Telephone interview — A structured telephone interview at three months will assess the degree of implementation, explore associated barriers (administrative, cognitive, organizational, ...), and investigate any potential link with hospital readmissions or changes in patients' living situations.

SUMMARY:
This single-center, prospective, observational cohort study aims to evaluate the actual implementation rate of social recommendations formulated by the Mobile Geriatric Team at Saint-Étienne University Hospital three months after hospital discharge. These recommendations may include human assistance, technical aids, financial aid applications, legal protective measures, or referrals to appropriate care structures.

A structured telephone interview at three months will assess the degree of implementation, explore associated barriers (administrative, cognitive, organizational, ...), and investigate any potential link with hospital readmissions or changes in patients' living situations.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 75 years or older
* Patients assessed by the Mobile Geriatric Team of the Saint-Etienne University Hospital with the formulation of social recommendations
* Patients residing at home or in a long-term care facility for dependent elderly individuals (nursing home / EHPAD)
* Informed consent obtained from the patient or their legal representative

Exclusion Criteria:

* Patients under 75 years old
* Refusal to participate in the study by the patient (or by the legally authorized representative/trusted person).
* Patients receiving exclusive palliative care
* Inability to ensure follow-up: in case of non-response at three months or in the event of death

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Any patient who has benefited from an assessment by the CHUSE EMG with formulation of social recommendations between August 1, 2025 and January 31, 2026 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Rate of implementation of social recommendations | Month : 3
  Evaluate the three-month implementation rate of the total social recommendations issued by the mobile geriatric team.

SECONDARY OUTCOMES:
Factors hindering the implementation of recommendations | Month : 3
  Identify the factors holding back the implementation of TOTAL recommendations (then SPECIFIC: human, technical, financial, patient orientation, implementation of legal protection measures).
Reasons for refusal or non-implementation | Month : 3
  Analyze the reasons for refusal or non-implementation.
Impact of non-implementation on the re-hospitalization rate | Month : 3
  Evaluate the impact of non-implementation on the re-hospitalization rate.
Patient's living environment | Month : 3
  Document changes in the patient's living environment at three months.

CONTACTS AND LOCATIONS:
Overall Officials: Manon SAHUC, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No